CLINICAL TRIAL: NCT06517108
Title: The Efficacy and Safety of Chuna Manual Treatment for Patients With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Chuna Manual Treatment for Patients With Primary Dysmenorrhea Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2021-18
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Primary Dysmenorrhea
Keywords: Chuna; Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chuna therapy (Experimental): 15 patients with chuna therapy
  Interventions: Procedure: Chuna therapy
- Physical therapy (Active Comparator): 15 patients with physical therapy
  Interventions: Procedure: Physical therapy

INTERVENTIONS:
Procedure: Chuna therapy — The chuna therapy group will receive chuna therapy based on the degree of displacement of the lumbar, ilium, sacrum, and cervical vertebrae. The type of weight or treatment is selected based on the clinical judgment of the Korean medicine practitioner (HVLA: high-velocity low-amplitude thrust, drop table manipulation, muscle energy techniques, myofascial release, etc.). The area and number of treatments performed are recorded separately. Thermotherapy is applied as an adjuvant treatment.
  The treatment will be administered between MCD 8 and MCD 28, twice a week during the 1st and 2nd cycle. The number of treatments can be adjusted depending on the patient's menstrual cycle and degree of displacement.
  Arms: Chuna therapy
Procedure: Physical therapy — The physical therapy group will receive transcutaneous electrical nerve stimulation (TENS) for about 10 to 15 minutes, and the area and number of times it was administered will be recorded. Thermotherapy is applied as an adjuvant treatment, and the area and number of times it is applied are recorded separately.
  The treatment will be administered between MCD 8 and MCD 28, twice a week during the 1st and 2nd cycle. The number of treatments can be adjusted depending on the patient's menstrual cycle and degree of displacement.
  Arms: Physical therapy

SUMMARY:
This study is a randomized controlled trial that compares 30 patients with primary dysmenorrhea by assigning them in a 1:1 ratio between patients treated with a Chuna therapy strategy and patients treated with a strategy using physical therapy. The purpose of the study is to confirm the comparative effectiveness of Chuna therapy and physical therapy.

DETAILED DESCRIPTION:
Menstrual pain is known to be caused by increased tension in the uterine muscles and irregular contractions, and is experienced by 50% of women who menstruate. However, most people control pain with NSAIDs or hormones. Among non-pharmacological treatments, manual therapy is known to control menstrual pain by influencing pain perception and pain-related serological factors. Previous research results have shown that manual therapy using sacroiliac joint correction and high-speed, low-amplitude thrust techniques is effective for menstrual pain. However, there is still no randomized controlled study limited to Chuna therapy. Therefore, the investigators would like to conduct a randomized clinical study to determine the effectiveness and safety of Chuna therapy for primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose menstrual pain is NRS 5 or higher during the last 3 months due to primary dysmenorrhea
* Patients who are between 14 and 49 years of age
* Patients whose cycle has been regular between 21 and 40 days for the past 3 months
* Patients who agree to participate in clinical research and provide written test subject consent

Exclusion Criteria:

* Patients whose cause of menstrual pain is determined to be an organic problem (uterine fibroids, adenomyosis, endometriosis, etc.) rather than a primary cause.
* Patients who have taken oral contraceptives or other hormonal therapy within the past 3 months.
* Patients diagnosed with other chronic diseases (stroke, myocardial infarction, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.) that may interfere with the treatment effect or interpretation of results.
* Patients who are currently taking steroids, immunosuppressants, drugs for mental illness, or other drugs that may affect the results of the study.
* Patients for whom manual therapy is inappropriate or unsafe: history of lumbar fusion or pelvic girdle surgery, spinal fracture, or severe instability.
* Pregnant women, those planning to become pregnant within 6 months, and those planning to take hormones such as oral contraceptives.
* Patients who finished participating in another clinical study less than 1 month ago, or who plan to participate in another clinical study during the study participation and follow-up period within 6 months from the date of selection.
* Patients who find it difficult to fill out the consent form for research participation.
* Other cases where participation in clinical research is deemed difficult by the researcher.

Ages: 14 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Peak dysmenorrhea NRS during menstrual period | Screening day(Cycle -1), At the first visit of Cycle 1, 2, 3, 5 (each cycle is 28 days)
  The maximum pain intensity during menstruation will be assessed using the NRS. In the NRS, patients choose a number from 0 to 10 that best represents their current level of discomfort (0 being no pain and 10 being the worst pain imaginable).

SECONDARY OUTCOMES:
EuroQol Visual Analogue Scale, EQ-VAS | At the first visit of Cycle 1, 2, 3, 5 (each cycle is 28 days)
  This assessment tool helps to express how good or bad a patient's health status is by having the patient record the degree of health status they feel on a vertical 100mm line, with one end indicating the worst imaginable health state and the other end indicating the best imaginable health state.
Modified pain scale | At the first visit of Cycle 1, 2, 3, 5 (each cycle is 28 days)
  The modified pain scale is a scale that defines pain according to work loss and the need for analgesics. It is the sum of the number of days of pelvic pain and use of painkillers, each calculated from 0 to a maximum of 3.
Short Form McGill Pain Questionnaire, SF-MPQ | At the first visit of Cycle 1, 2, 3, 5 (each cycle is 28 days)
  The main component of the SF-MPQ consists of 15 words (11 sensations, 4 emotions) rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate, or 3 = severe. The three pain scores are obtained as the sum of the intensity values of the selected words. Also included is the current pain intensity (PPI) index and visual analog scale (VAS) from the standard MPQ. The Korean version of SF-MPQ, adapted by Kim Eun-ju, is used.
Positive and Negative Affect Schedule, PANAS | At the first visit of Cycle 1, 2, 3, 5 (each cycle is 28 days)
  The positive and negative emotion scales developed by Watson et al. consist of a total of 20 questions, including 10 positive emotion scales and 10 negative emotion scales. Evaluate the degree to which each item applies to you on a 5-point scale (0 = not at all, 1 = slightly, 2 = moderately, 3 = a lot, 4 = very much).
EuroQol-5 Dimension, EQ-5D-5L | At the first visit of Cycle 1, 2, 3, 5 (each cycle is 28 days)
  It is the most widely used of several indirect measurement methods as a method of indirectly calculating the quality weight of a specific health state using pre-assigned preference scores for each functional level after evaluating the health state from various aspects. The EQ-5D-5L consists of 5 questions. Each question includes mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Ask about the degree of depression, etc. Each item is weighted according to its level, and an equation for calculating preference scores is presented based on these weights and constants.
Short Form-12 Health Survey version 2, SF-12 v2 | At the first visit of Cycle 1, 2, 3, 5 (each cycle is 28 days)
  Health-related quality of life (HRQoL) The evaluation questionnaire consists of 12 questions spanning 8 areas (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health). It usually takes less than 5 minutes to complete, and higher scores indicate better health-related quality of life. SF-12 is used to evaluate the functional health and well-being of patients and healthy people.
Patient Global Impression of Change, PGIC | At the first visit of Cycle 3, 5 (each cycle is 28 days)
  This is a method that allows the patient to subjectively evaluate the degree of improvement on a 7-level scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Sunah Kim, KMD, Principal Investigator — Daejeon Jaseng Hospital of Korean Medicine
Locations (1):
- Daejeon Jaseng Hospital of Korean Medicine, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No